CLINICAL TRIAL: NCT05343403
Title: Collaborating to Improve Neonatal Care: ParentAl paRticipation on The NEonatal waRd - the neoPARTNER Study
Brief Title: Parental Participation on the Neonatal Ward - the neoPARTNER Study
Acronym: neoPARTNER
Status: Active, not recruiting | Type: Observational
Sponsor: Onze Lieve Vrouwe Gasthuis (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Dr. Sophie van der Schoor, Principal Investigator, Onze Lieve Vrouwe Gasthuis
Other Study IDs: NL78176.100.21
Record Dates: First submitted 2022-02-16; First posted 2022-04-25 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Premature; Premature Birth; Prematurity; Perinatal Problems; Neonatal Sepsis; Neonatal Infection; Neonatal Hyperbilirubinemia; Infant Development; Infant, Newborn, Disease; Infant, Premature, Diseases; Infant, Small for Gestational Age; Small for Gestational Age Infant; Maternal Distress; Parent-Child Relations; Parents
Keywords: Family Centred Rounds; Family Integrated Care; Shared Decision Making; Parent participation
MeSH Terms: conditions — Premature Birth; Neonatal Sepsis; Hyperbilirubinemia, Neonatal; Disease; Infant, Premature, Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — saliva, buccal mucosa, hair, human's milk
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Family Integrated Care: During the intervention period, Family Integrated Care (FICare) will be implemented on the neonatal wards of the participating hospitals. Families that are included during this intervention period will participate in Family Centred Rounds (FCR), while being supported by the principles of FICare. FICare incorporates psychological, educational, communication, and environmental strategies to support parents and to prepare them emotionally, cognitively, and physically to care autonomously for their infant at the time of discharge. In FCR, parents actively participate in the medical rounds and decisions are made based on shared-decision making. Not only are parents informed about the clinical condition of their child, they can ask questions and share their own valuable information on their child. Such information can include the overall wellbeing but also specific medical information.
  Interventions: Other: Family Integrated Care
- Standard Neonatal Care: In the control period, standard neonatal care (SNC) will be provided. Medical rounds will be held between healthcare professionals, and parents are not (structurally) participating during these rounds. Parents are updated daily by the nurses, and (usually) weekly by their attending physician. Care for the infants is provided mostly by the nurses. Parents usually have (unlimited) access to the ward, but are not supported by the concept of FICare. As such, they do not receive education and are not structurally supported by veteran parents. Healthcare professionals stimulate parents to participate in daily care (such as feedings or skin-to-skin care), but do not receive structural education on how to incorporate parents as equal partners into the care team.

INTERVENTIONS:
Other: Family Integrated Care — The intervention will consist of FICare, including parental participation in medical rounds (FCR). Parents and healthcare professionals will be educated and supported by the four pillars of FICare: parent education, education of healthcare professionals, psychosocial support and a supportive environment of the neonatal ward.
  Groups: Family Integrated Care

SUMMARY:
Objective: To investigate the effect of FCR as part of the FICare principles during hospital stay, on parental stress at discharge in parents of preterm or ill infants admitted to the neonatal ward for >7 days as compared to standard medical rounds (SMR) without parents as part of standard neonatal care (SNC).

DETAILED DESCRIPTION:
Parents are often appointed a passive role during the admission of their preterm (born before 37 weeks of gestational age) or illinfant. Multiple studies have demonstrated that information and communication are crucial for families of intensive care patients.However, common practice in neonatal wards regarding daily rounds is that the medical rounds are only attended by the physicianand nurse without presence and participation of the parents. Parents are usually updated by the nurse afterwards. Family CentredRounds (FCR) include parents on daily rounds (digital or physical presence), involving them in the process of patient management,allowing them to hear their infants' conditions first-hand, to provide information on their child's general wellbeing themselves and toask questions and participate in shared decision making. Family Integrated Care (FICare) comprises a framework to implement FCRby bringing parents, medical and nursing staff together and involving parents as equal partners, minimizing separation, andsupporting parent-infant closeness. FICare consists of a collaborative program of psychological, educational, communication, andenvironmental strategies to support parents to cope with neonatatal environment and to prepare them to be able to emotionally,cognitively, and physically care for their infant.

Objective of the study: To investigate the effect of FCR during hospital stay, accompanied by FICare, on parental stress at discharge in parents of preterm(born before 37 weeks of gestational age) or ill (for instance with sepsis or small for gestational age) infants admitted to the neonatalward for >7 days as compared to standard daily rounds (SDR) without parents with SNC. We primarily hypothesize that FCR andFICare are superior to SNC with regard to parental stress at discharge. Secondary outcomes in parents include participation inneonatal care, experience in shared decision making, parent-infant bonding, biomarkers of stress (in hair and saliva), breastmilkcomposition and the longitudinal course of parent mental health after infant discharge. Infant outcomes include breastfeeding atdischarge, growth, biomarkers of stress in saliva and length of hospital stay. For healthcare professionals outcomes such as workengagement and autonomy will be analysed at the cluster level. Cost-effectiveness analysis will be done as well at the level ofparents and healthcare professionals.

Study design: A multicentre stepped wedge cluster randomised trial will be conducted. A total of 10 hospitals with a level 2 neonatal ward in theNetherlands will participate. Timing of start of intervention will be randomised between sites.

Study population: All (parents of) infants admitted to the neonatal ward directly after birth, or transferred to a participating centre after birth in aneonatal intensive care unit (NICU) are eligible for participation in the study.

Intervention (if applicable): The intervention will consist of parental participation in medical rounds (FCR). Parents and healthcare professionals will besupported by the four pillars of FICare: parent education, education of healthcare professionals, psychosocial support andenvironment of the neonatal ward.

Primary study parameters/outcome of the study: The main outcome is parental stress at discharge, as defined by the total score on the Parental Stress Scale (PSS:NICU). ThePSS:NICU is a three-dimensional tool, in which parents express the amount of stress they experienced by rating 26 items on a 5-point Likert scale ("not stressful at all" to "extremely stressful").

Secundary study parameters/outcome of the study (if applicable): Secondary outcome measures on the individual level will be parent participation in neonatal care, parent-infant bonding andexperiences in shared decision making. The longitudinal course of parental mental health (anxiety, depression, posttraumatic stress)will be analyzed, as well as biomarkers of stress (in saliva, hair and breastmilk) and breastmilk composition. Also, neonatalsecondary outcome measures will be taken into account, specifically length of stay, breastfeeding rates at discharge, biomarkers ofstress in saliva and growth. On the cluster level we will study professional secondary outcome measures such as work engagementand autonomy.

ELIGIBILITY:
Inclusion Criteria:

* Infant requiring hospital admission directly (within 24 hours) after birth;
* Parent of 18 years or older;
* Written informed consent of both parents.

Exclusion Criteria:

* Infant's hospital stay shorter than 7 days;
* Infant with severe congenital or syndromal anomaly;
* Infant with critical illness who is unlikely to survive;
* Parent with current psychosocial problems (such as posttraumatic stress disorder, schizophrenia or psychotic disorders) with or without medication which have not been stable over the past year;
* Involvement of child protective services in the family;
* Parent not able or not willing to fill out questionnaires in English or Dutch.

Min Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A total of 600 preterm or ill infants, admitted 37 days to a level 2 neonatal ward, with their parents (600 mothers and 600 fathers/partners) will be included in this study.
  Moreover, healthcare professionals working at the different hospitals will be included as well.
Sampling Method: Probability Sample
Enrollment: 613 (Actual)
Dates: Start 2022-03-07 (Actual); Primary Completion 2024-02-02 (Actual); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Level of parental stress | Immediately after intervention (at discharge of the infant)
  Patient Reported Outcome: Parental Stress Scale: Neonatal Intensive Care Unit (Miles, 1993). Range: 0-135 points, higher score indicating higher levels of parental stress.

SECONDARY OUTCOMES:
Experiences of Shared Decision Making | Immediately after intervention (at discharge of the infant)
  Patient Reported Outcome: Shared Decision Making Questionnaire (SDM-Q-9, Kriston et al. 2010). Range: original score of 0-45 points calculated into score with range of 0-100 points, higher score indicating higher levels of shared decision making.
Parent-infant attachment | Immediately after intervention (at discharge of the infant)
  Maternal (or Paternal) Postnatal Attachment Scale (Condon et al., 1998). Range: 19-95 points, lower score indicating problematic mother-to-infant bonding or father-to-infant bonding, respectively.
Level of parental participation in neonatal care | Immediately after intervention (at discharge of the infant)
  Patient Reported Outcome: CO-PARTNER tool (van Veenendaal et al, 2021). Range: 0-62, higher score indicating higher level of participation.
Symptoms of parental depression | Pre- and post-intervention, measured at discharge of the infant through study completion at the (corrected) age of 12 months
  Patient Reported Outcome: PROMIS Depression, Shortform (PROMIS Health Organisation). Range: 8-40 points (calculated into a T-score with a mean of 50 and a standard deviation of 10), higher score indicating more symptoms of depression.
Symptoms of parental anxiety | Pre- and post-intervention, measured at discharge of the infant through study completion at the (corrected) age of 12 months, 3, 6 and 12 months corrected age
  Patient Reported Outcome: PROMIS Anxiety, Shortform (PROMIS Health Organisation). Range: 8-40 points (calculated into a T-score with a mean of 50 and a standard deviation of 10), higher score indicating more symptoms of anxiety.
Symptoms of parental posttraumatic stress | Pre- and post-intervention, measured at discharge of the infant through study completion at the (corrected) age of 12 months
  Patient Reported Outcome: Post-traumatic Stress Disorder Checklist for DSM-5 (Weathers et al., 2013). Range: 0-80, higher score indicating more symptoms of posttraumatic stress.
Cost-effectiveness on parent and infant level | At the corrected age of 12 months.
  Patient Reported Outcome: Productivity Cost Questionnaire & Medical Consumption Questionnaire (Bouwmans et al, 2015 & 2013, respectively). No scale applicable.
Infant development | At the corrected age of 12 months.
  Patient Reported Outcome: Ages and Stages Questionnaire, edition 3 (Flamant et al, 2011). Range: 0-300 points, higher score indicating better infant development.
Length of hospital stay (infant) | During intervention (estimated average of 21 days).
  Duration of the hospital admission of the infant, expressed in days.
Amount of breastfeeding | Immediately after intervention (at discharge of the infant).
  Amount of breastfeeding defined as percentage of total (enteral) intake
Infant growth | Pre- and post-intervention, measured at discharge of the infant through study completion at the (corrected) age of 12 months
  Rate of weight gain during hospital stay and during first year of life.
Change in experience of Shared decision making (healthcare professionals) | Through study completion, an average of 21 months.
  Self-reported outcome: Shared Decision Making Questionnaire-Physician Version. (Rodenburg-Vandenbussche et al., 2015). Range: original score of 0-45 points calculated into score with range of 0-100 points, higher score indicating higher levels of shared decision making.
Change in experienced work engagement (healthcare professionals) | Through study completion, an average of 21 months.
  Self-reported outcome: Utrechtse Work Engagement Scale (Schaufeli et al., 2003). Range: 0-6 points, higher score indicating higher levels of work engagement.
Change in experienced work autonomy (healthcare professionals) | Through study completion, an average of 21 months.
  Self-reported outcome: Job Content Questionnaire, Decision Authority Subscale (Karasek et al., 1998). Range: 3-12 points, higher score indicating more feeling of autonomy.
Cost-effectiveness (healthcare professionals) | Through study completion, an average of 21 months.
  Work absence as registered at the hospital administration, and self-reported outcome: Productivity Cost Questionnaire (Bouwmans et al., 2015). No range applicable.
Family Centred Rounds | Through study completion, an average of 21 months.
  % of medical rounds with parental presence as reported by healthcare professionals

CONTACTS AND LOCATIONS:
Overall Officials: Sophie van der Schoor, Dr., Principal Investigator — OLVG
Locations (10):
- Netherlands (10):
  - Flevoziekenhuis, Almere Stad, Flevoland
  - Amphia Ziekenhuis, Breda, North Brabant
  - Noordwest Ziekenhuisgroep, Alkmaar, North Holland
  - Ziekenhuis Amstelland, Amstelveen, North Holland
  - BovenIJ Ziekenhuis, Amsterdam, North Holland
  - Tergooi Medisch Centrum, Blaricum, North Holland
  - Zaans Medisch Centrum, Zaandam, North Holland
  - Medisch Spectrum Twente, Enschede, Overijssel
  - Franciscus Gasthuis & Vlietland, Rotterdam, South Holland
  - Juliana Kinderziekenhuis, The Hague, South Holland

REFERENCES:
- [Background] Hoeben H, Alferink MT, van Kempen AAMW, van Goudoever JB, van Veenendaal NR, van der Schoor SRD, On Behalf Of The neoPARTNER Study Group. Collaborating to Improve Neonatal Care: ParentAl Participation on the NEonatal Ward-Study Protocol of the neoPARTNER Study. Children (Basel). 2023 Aug 30;10(9):1482. doi: 10.3390/children10091482. PMID 37761442
- [Derived] Alferink MT, Hoeben H, Jonkman NH, van Goudoever JB, van Kempen AAMW, van Veenendaal NR, van der Schoor SRD; neoPARTNER studygroup. Family integrated care reduces stress in transferred parents of preterm infants, but not across all families: a stepped-wedge cluster-randomized trial. J Perinatol. 2025 Jun;45(6):797-805. doi: 10.1038/s41372-025-02318-w. Epub 2025 May 20. PMID 40394238